CLINICAL TRIAL: NCT05381818
Title: Preoperative Inspiratory Muscle Strength Training and Pulmonary Complications After Surgery
Brief Title: Pre-operative Inspiratory Muscle Strength Training in Total Joint Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB202102681; R21AG083667 (NIH)
Record Dates: First submitted 2022-05-16; First posted 2022-05-19 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Arthropathy of Knee; Arthropathy of Hip; Lower Extremity Fracture; Orthopedic Disorder
Keywords: Inspiratory muscle training; Pulmonary complications; Total joint replacement
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Daily IMT (dIMT) (Experimental): IMT (inspiratory muscle training) is a treatment strategy aimed to strengthen the muscles of inspiration, the diaphragm and external intercostals, by increasing their force-generating capacity. Participants in the dIMT (daily IMT) will complete daily inspiratory training exercises 2-4 weeks prior to surgery. A pressure threshold training device containing an adjustable-tension spring to provide resistance during inspiration will be used. Subjects will complete 5 sets of 5 maximal volume and speed breaths daily at a pressure 70% of MIP and will rest 1 minute between sets. They will be asked to keep a log to track their sessions to evaluate compliance with the exercise regimen.
  Interventions: Behavioral: Daily Inspiratory Muscle Training (dIMT)
- Acute IMT (aIMT) (Active Comparator): Patients in the aIMT (acute IMT) experimental group will complete a single session of IMT guided by a physical therapist within 30 minutes of anesthesia induction in addition to standard of care. The adjustable pressure threshold training device to provide resistance during inspiration will be used. Subjects will complete 5 sets of 5 maximal volume and speed breaths, and rest 1 minute between sets. The training intensity will be set at 70% of MIP.
  Interventions: Behavioral: Acute Inspiratory Muscle Training (aIMT)
- Standard of Care (SOC) (Active Comparator): The SOC group will receive the usual surgical standard of care only.
  Interventions: Other: Standard of Care (SOC)

INTERVENTIONS:
Behavioral: Daily Inspiratory Muscle Training (dIMT) — Daily IMT training sessions for 2-4 weeks prior to surgery
  Arms: Daily IMT (dIMT)
Behavioral: Acute Inspiratory Muscle Training (aIMT) — A single session of IMT provided within 30 minutes prior to anesthesia induction.
  Arms: Acute IMT (aIMT)
Other: Standard of Care (SOC) — Standard of care only pre and post-operatively.
  Arms: Standard of Care (SOC)

SUMMARY:
The purpose of this research study is to evaluate effects of respiratory strengthening exercises on breathing function, in people who have orthopedic surgery. It is known that breathing function decreases for a few days after surgery. in In this study, we want to see if exercising before surgery strengthens the breathing muscles and improves recovery after surgery.

DETAILED DESCRIPTION:
Preoperative inspiratory muscle training (IMT) has been shown to reduce post operative complications (PPC's) following prolonged cardiac surgeries, but its potential benefits have not been investigated in shorter surgeries with expected brief post-operative hospitalizations. We intend to address this unmet need by investigating preoperative IMT, an evidence-based rehab strategy to optimize lung function, prior to total joint arthroplasty surgery. The fundamental hypothesis guiding this proposal is that preoperative IMT will attenuate post-operative declines in breathing function and offset PPCs. To test this hypothesis, we will conduct a single center, randomized, prospective pilot study. Adults scheduled for total joint arthroplasty or lower extremity orthopedic surgery will be randomized to either complete daily IMT in advance of surgery (dIMT), a single acute IMT session immediately before surgery (aIMT), or usual surgical standard of care (SOC). Inspiratory muscle strength and pulmonary function will be evaluated upon enrollment ~4 weeks in advance of surgery and in pre-operative holding, and post-operative declines will be investigated through the first 24 hours (Aim 1). Further, we will investigate the effect of training assignment on post-operative clinical outcomes (Aim 2).

ELIGIBILITY:
Inclusion Criteria:

* 18 or older
* History of current or previous tobacco use (including vaping containing nicotine products)
* One or more risk factors for post operative pulmonary complications including history of current or previous tobacco use, a clinically diagnosed lung disease, shortness of breath with minimal exertion, FEV1 or FVC less than 80% than predicted or respiratory muscles strength below lower limit of normal for age and sex.
* History of smoking related lung disease
* Projected surgical time > 30 minutes
* Ability to follow instructions to complete IMT exercises
* Ability to communicate adverse effects such as pain or fatigue or the need for assistance

Exclusion Criteria:

* American Society of Anesthesiologists physical status classification of 4 or greater .
* Recent history of acute pneumonia or lower respiratory infection in the previous two weeks requiring acute corticosteroid or antibiotic medication,
* Preoperative dependence on continuous supplemental oxygen dependence.
* Preoperative dependence on positive pressure breathing support while awake and upright (night time CPAP permitted),
* Diagnosis of a neurologic condition (i.e. MS, ALS, Parkinson's, stroke),
* Participating in a pulmonary rehabilitation program
* Severe obstructive pulmonary disease (Classification of Global Initiative for Chronic Obstructive Lung Disease (GOLD) 3 or higher, indicating FEV1<50% predicted.
* Patients with an infectious disease requiring isolation (i.e. COVID-19).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Maximal Inspiratory Pressure (MIP) | 24-hours post-op.
  Measure of strength of inspiratory muscles.
Forced vital capacity (FVC) | 24-hours postoperative changes
  The volume of air that can be forcefully exhaled after a full inhalation.

SECONDARY OUTCOMES:
Post operative pulmonary complications | 10 days Post-op
  Incidence of post-operative pulmonary complications

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Smith, PhD, Principal Investigator — University of Florida, College of Public Health and Health Professions - Gainesville
Locations (1):
- University of Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No